CLINICAL TRIAL: NCT00017056
Title: A Phase II Study Of Epothilone Analog BMS-247550 In Patients With Metastatic Gastric Adenocarcinoma Previously Treated With A Fluoropyrimidine And/Or Platinum
Brief Title: BMS-247550 in Treating Patients With Recurrent Metastatic Stomach Cancer That Has Been Previously Treated With Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 01-015; CDR0000068645 (Registry Identifier: PDQ (Physician Data Query)); NCI-G01-1950
Record Dates: First submitted 2001-06-06; First posted 2004-02-16 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage IV gastric cancer; recurrent gastric cancer; stage IV esophageal cancer; recurrent esophageal cancer; adenocarcinoma of the stomach; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — ixabepilone

INTERVENTIONS:
Drug: ixabepilone

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of BMS-247550 in treating patients who have recurrent metastatic stomach cancer that has been previously treated with chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the clinical activity of BMS-247550 in terms of response rate in patients with recurrent metastatic gastric cancer previously treated with a fluoropyrimidine or platinum regimen. II. Determine the safety of this drug in this patient population. III. Determine the duration of response, time to progression, and survival of patients treated with this drug.

OUTLINE: This is a multicenter study. Patients receive BMS-247550 IV over 1 hour on day 1. Treatment repeats every 21 days for up to 18 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive up to 4 additional courses after CR. Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 21-58 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent metastatic adenocarcinoma of the stomach or gastroesophageal junction No squamous cell or sarcomatous elements in tumor Previously treated with 1 prior fluoropyrimidine and/or platinum based chemotherapy regimen for metastatic disease OR Recurrent disease within 6 months of completing adjuvant fluoropyrimidine-containing therapy Bidimensionally measurable disease No known brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 2,000/mm3 Platelet count greater than 125,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) ALT no greater than 2.5 times ULN (5 times ULN if liver metastases present) Renal: Creatinine no greater than 2 times ULN Cardiovascular: No unstable angina, myocardial infarction, or congestive heart failure within the past 6 months Other: No grade 2 or greater neuropathy (motor or sensory) No other malignancy within the past 2 years except nonmelanoma skin cancer or carcinoma in situ of the cervix No serious concurrent infection No other medical illness that would preclude study No psychiatric disorder or other condition that would preclude study No known hypersensitivity to Cremophor EL Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 2 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Chemotherapy: See Disease Characteristics At least 3 weeks since prior chemotherapy Prior adjuvant or neoadjuvant chemotherapy allowed No more than 1 prior chemotherapy regimen for metastatic disease No prior taxane therapy No other concurrent chemotherapy Endocrine therapy: No concurrent hormonal therapy except hormone replacement therapy Radiotherapy: At least 3 weeks since prior radiotherapy and recovered No prior radiotherapy to major bone marrow-containing areas (pelvis, lumbar spine) or to only site of measurable disease No concurrent therapeutic radiotherapy Surgery: At least 1 week since prior minor surgery and recovered At least 3 weeks since prior major surgery and recovered Other: No other concurrent experimental anticancer medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-02; Primary Completion 2002-01 (Actual); Study Completion 2002-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manish A. Shah, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States